CLINICAL TRIAL: NCT05720819
Title: Utility of a Novel, Combined Biofeedback-Virtual Reality Device as Adjunctive Treatment for Chronic Migraine
Brief Title: Biofeedback-VR for Treatment of Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ami Cuneo, Acting Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010685
Record Dates: First submitted 2022-12-21; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Chronic Migraine; Behavioral Treatment; Biofeedback; Virtual Reality; Medication Overuse Headache
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Intervention Model Description: This study is a randomized, pilot study comparing the intervention of combined biofeedback-VR plus standard medical care as treatment for chronic migraine versus a wait-list control group receiving standard medical care alone as treatment for chronic migraine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Biofeedback-VR intervention plus standard clinical care) (Experimental): This arm includes individuals with chronic migraine receiving the home-based biofeedback-VR intervention plus standard medical care as treatment for chronic migraine
  Interventions: Device: Combined biofeedback-virtual reality device
- Control Group (standard clinical care alone) (No Intervention): This arm, a wait-list control group, includes individuals with chronic migraine receiving standard medical care alone as treatment for chronic migraine.

INTERVENTIONS:
Device: Combined biofeedback-virtual reality device — The study's biofeedback-VR device was developed in collaboration with students and faculty at the University of Washington Global Innovation Exchange program. The system included an Oculus Go mobile VR headset (wireless, portable, head-mounted display, with screen providing a 101° field of view with 2560 x 1440 resolution at a 60-72 Hz frame rate; Oculus VR, LLC, Menlo Park, CA/USA) and with built-in speaker, in addition to a Polar H10 heart rate monitor (electrocardiogram, or ECG, to measure heart rate; Polar Electro Inc., Bethpage, NY/USA), with customized software programmed for the study using the Unity3D game engine (Unity Technologies, Bellevue, WA/USA). Individuals in the experimental arm are asked to use this device for 10 minutes daily, on at least 3 days per week.
  Arms: Intervention Group (Biofeedback-VR intervention plus standard clinical care)

SUMMARY:
Migraine is a common, debilitating neurologic condition affecting more than 900 million individuals worldwide. Established treatments for migraine include medications, vitamin and herbal supplements, neuromodulation, and behavioral treatment strategies. This study aims to determine whether a novel, home-based behavioral approach, combined biofeedback-virtual reality therapy, can improve self-reported migraine-related outcomes in individuals living with chronic migraine.

In this randomized, controlled pilot study, 50 adults with chronic migraine are randomized to the experimental group (frequent use of a heart rate variability biofeedback-virtual reality device plus standard medical care; n=25) or wait-list control group (standard medical care alone; n=25). The primary outcome is reduction in mean monthly headache days between groups at 12 weeks. Secondary outcomes include mean change in acute analgesic use frequency, depression, migraine-related disability, stress, insomnia, and catastrophizing between groups at 12 weeks. Tertiary outcomes include change in heart rate variability and device-related user experience measures.

DETAILED DESCRIPTION:
Chronic migraine (CM) is a debilitating neurologic condition affecting 1-2% of the population. By definition, individuals with CM experience at least 15 headache days per month (including at least 8 migraine days) for more than 3 months. In addition to frequent, debilitating headaches, CM is associated with increased rates of headache-related disability, psychiatric comorbidity, pain catastrophizing, insomnia, risk of medication overuse headache, and healthcare resource utilization.

Established treatments for migraine include medications, vitamin and herbal supplements, neuromodulation, and behavioral treatment strategies. Our study aims to determine whether a novel, home-based behavioral approach, combined biofeedback-virtual reality therapy, can improve self-reported migraine-related outcomes in individuals living with chronic migraine.

In this randomized, controlled pilot study, 50 adults with chronic migraine are randomized to the experimental group (frequent use of a heart rate variability biofeedback-virtual reality device plus standard medical care; n=25) or wait-list control group (standard medical care alone; n=25). The primary outcome is reduction in mean monthly headache days between groups at 12 weeks. Secondary outcomes include mean change in acute analgesic use frequency, depression, migraine-related disability, stress, insomnia, and catastrophizing between groups at 12 weeks. Tertiary outcomes include change in heart rate variability and device-related user experience measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of International Classification of Headache Disorders (ICDH-3 beta) criteria for chronic migraine
* Individuals having experienced least 15 headache days per month (including at least 8 migraine days per month) in the preceding 3 months
* Ability to speak English or Spanish

Exclusion Criteria:

* Individuals with cognitive impairment, severe psychiatric comorbidities (including active suicidal or homicidal ideation and/or psychosis), hearing/seeing difficulties, epileptic or non-epileptic seizures, and prisoners.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Mean headache days per month | Baseline compared with week 12
  Mean headache days per month in the experimental group, as compared with mean headache days per month in the control group.

SECONDARY OUTCOMES:
Frequency of total acute analgesic medication uses per month | Baseline compared with week 12
  Frequency of total acute analgesic medication uses per month in the experimental group, as compared with total acute analgesic medication uses per month in the control group.
Depression score (Patient Health Questionnaire-8) | Baseline compared with week 12
  Depression score in the experimental group, as compared with depression score in the control group. The lowest attainable score is 0 and the highest attainable score is 24. A score of 0-4 is no depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-24 severe depression.
Migraine associated disability score (Migraine Disability Assessment) | Baseline compared with week 12
  Migraine associated disability score in the experimental group, as compared with the migraine associated disability score in the control group. Minimum score is 0, maximum score is indefinite. Score of 0-5 is defined as minimal disability, 6-10 as mild disability, 11-20 as moderate disability, and score of at least 21 is severe disability.
Stress score (Perceived Stress Scale) | Baseline compared with week 12
  Stress score in the experimental group, as compared with the stress score in the control group. Minimum score is 0, maximum score is 40. Score 0-13 is low stress, 14-26 reflects moderate stress, 27-40 reflects high stress.
Catastrophizing score (Concerns about Pain scale) | Baseline compared with week 12
  Catastrophizing score in the experimental group, as compared with the catastrophizing score in the control group. The minimum score is 6 and the maximum score is 30. Scores are converted into a T score metric. A higher score suggests increased concern about pain.

OTHER OUTCOMES:
Heart rate variability score | Baseline compared with week 12
  Measurement of average heart rate variability in the experimental group alone.
Qualitative impressions of the intervention | Baseline compared with week 12
  Qualitative impressions of experience with the biofeedback-virtual reality treatment for the experimental group alone. This is measured via questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Ami Z Cuneo, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No